CLINICAL TRIAL: NCT06431360
Title: Effect of Strontium-90 Brachytherapy Combined With Hyperthermia in the Treatment of Keloid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Director of nuclear medicine department, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20240514-02
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — Diathermy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Sr-90 brachytherapy followed by hyperthermia.
  Interventions: Other: hyperthermia
- Control group (No Intervention): Sr-90 brachytherapy alone.

INTERVENTIONS:
Other: hyperthermia — hyperthermia (using a heater, 44℃for 15 min)
  Other Names: heater
  Arms: Experimental group

SUMMARY:
Keloid patients were randomized into the experimental and control groups. Experimental group: Strontium-90 (Sr-90) brachytherapy followed by hyperthermia. Control group: Sr-90 brachytherapy alone .

DETAILED DESCRIPTION:
Sr-90 brachytherapy: 6-7 Gy each time, twice a week for 3 weeks; Hyperthermia: using a heater, 44℃ for 15 min

ELIGIBILITY:
Inclusion Criteria:

* The patient was clinically diagnosed with keloid, and the keloid area was clean without rupture and exudation；
* Body surface keloid thickness: 2~5mm, diameter ≥10mm.

Exclusion Criteria:

* Women who plan to become pregnant within 3 months or are pregnant or breastfeeding;
* Patients with cicatricial constitution;
* Abnormal coagulation function;
* Patients who have received an adequate dose or course of radiation therapy;
* People with previous immune system diseases, diabetes and other metabolic diseases.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) scores | once every 3 months for 1 year after the last treatment
  The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability and surface area). All items are scored on a scale ranging from 1 ('like normal skin') to 10 ('worst scar imaginable'). The sum of the six items results in a total score of the POSAS observer scale. Categories boxes are added for each item. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.
  comparable anatomic location.
Vancouver Scar Scale (VSS) scores | once every 3 months for 1 year after the last treatment
  Physician evaluation comprised the use of the Vancouver Scar Scale (VSS) to evaluate the pigmentation (0=normal, 1=hypopigmented, 2=hyperpigmented), pliability (0=normal, 1= supple, 2=yielding, 3=firm, 4=banding, 5=contracture), height (0= flat, 1=5 mm), and vascularity (0=normal, 1=pink, 2=pink to red, 3=red, 4=red to purple, 5=purple).

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Study Director — Nanjing First Hospital, Nanjing Medical University
Locations (2):
- China (2):
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical Univerity, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No